CLINICAL TRIAL: NCT02605369
Title: SURVIVAL PLUSS: Increasing Capacity for Mama-baby Survival in Post-conflict Uganda and South Sudan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Makerere University (Other)
Collaborators: Centre For International Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015-121
Record Dates: First submitted 2015-11-12; First posted 2015-11-16 (Estimated); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Neonatal Death; Preterm Birth; Low Birthweight; Neonatal Hypoglycemia
Keywords: Facility births
MeSH Terms: conditions — Perinatal Death; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm: An integrated package (Experimental): Pregnant women in the intervention clusters will receive an integrated package consisting of peer support for facility based births by pregnancy buddies, mama kits and mobile phone messages. These components will all aim at mitigating the three delays and increasing the proportion of facility based births.
  Interventions: Behavioral: Intervention arm: An integrated package
- Control arm: Standard of care (No Intervention): Pregnant women in the control clusters will continue to receive the standard of care for pregnant women according to Ugandan Ministry of Health guidelines

INTERVENTIONS:
Behavioral: Intervention arm: An integrated package — See description in previous column
  Arms: Intervention arm: An integrated package

SUMMARY:
Universal coverage of good quality facility based care globally could prevent nearly 113,000 maternal deaths, 531,000 stillbirths and 1.3 million neonatal deaths annually by 2020. Yet, only 57% of pregnant Ugandan women choose to deliver at health facilities. This unacceptably low coverage of facility based births could explain, in part, the high maternal and perinatal mortality estimates in Uganda. While multiple studies have examined factors associated with this low utilization of health services around the time of birth, there is inadequate implementation research exploring the best systematic methods that could promote uptake and scale up of facility based births. This study will therefore examine the effect of an intervention package (peer counselling by pregnancy buddies on facility based births, mobile phone messaging promoting facility based births and provision of mama-kits) on the frequency of facility based births and perinatal mortality. The study, a cluster randomized community based intervention trial in post-conflict Northern Uganda, will provide data crucial in framing national policy regarding measures to promote the use of health facilities.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women at 28 or more weeks of gestation
* Residence in the selected clusters
* Pregnant women under 18 years of age will be included since they are considered as emancipated minors in Uganda

Exclusion Criteria:

* Intention to move from the study area within one year
* Psychiatric ailments that may inhibit the informed consent process

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1877 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Facility based birth | Day 1
  Delivery at a health facility

SECONDARY OUTCOMES:
Neonatal death | Day 28
  Death within the first month of life
Timely initiation of breastfeeding | Up-to one hour after birth
  Initiation of breastfeeding with the first hour after birth
Severe illness | Day 28
  Severe illness within the first month of life
The percent of newborns attended by a health care pro-vider during the first 48 hours following birth | Up-to 48 hours after birth
  Proportion of babies seen by a health care work in the first 48 hours after birth
The percent of newborns attended by a health care pro-vider during the first 7 days following birth | 1 week
  Proportion of babies seen by a health care work in the first one week after birth

OTHER OUTCOMES:
Low birthweight | Up-to 48 hours after birth
  Proportion of infants with a birthweight =< 2500gms
Preterm birth | 7 days postpartum
  Proportion of infants born at less than 37 completed weeks of gestation measured by the New Ballad Score
Neonatal hypoglycemia | Up-to 7 days after birth
  Proportion of infants with random blood glucose less than 47mg/dl

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Nankabirwa, MD, MPH, PhD, Principal Investigator — Department of Epidemiology and Biostatistics, School of Public Health, College of Health Sciences, Makerere University; James K Tumwine, MD, PhD, Principal Investigator — Makerere University; Grace Ndeezi, MD, PhD, Principal Investigator — Makerere Univeristy; Thorkild Tylleskar, MD, PhD, Principal Investigator — University of Bergen; Paul Wako, MD, PhD, Principal Investigator — Busitema University; Joyce Kaducu, Principal Investigator — Gulu University; Jino Meleby, Principal Investigator — University of Juba; Frederik Froen, MD, PhD, Principal Investigator — Norwegian Institute of Public Health
Locations (1):
- Lira District, Lira, Uganda

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and/or analyzed during the current study will be available on reasonable request

REFERENCES:
- [Derived] Nankabirwa V, Mukunya D, Ndeezi G, Odongkara B, Arach AA, Achora V, Mugenyi L, Sebit MB, Wandabwa JN, Waako P, Tylleskar T, Tumwine JK. Can an integrated intervention package including peer support increase the proportion of health facility births? A cluster randomised controlled trial in Northern Uganda. BMJ Open. 2024 Feb 7;14(2):e070798. doi: 10.1136/bmjopen-2022-070798. PMID 38326267
- [Derived] Mukunya D, Tumwine JK, Nankabirwa V, Odongkara B, Tongun JB, Arach AA, Tumuhamye J, Napyo A, Zalwango V, Achora V, Musaba MW, Ndeezi G, Tylleskar T. Neonatal hypothermia in Northern Uganda: a community-based cross-sectional study. BMJ Open. 2021 Feb 11;11(2):e041723. doi: 10.1136/bmjopen-2020-041723. PMID 33574146